CLINICAL TRIAL: NCT01183104
Title: Efficacy and Safety Comparison of Sitagliptin and Glimepiride in Elderly Japanese Patients With Type 2 Diabetes
Brief Title: START-J: SiTAgliptin in eldeRly Trial in Japan
Acronym: START-J
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Japan Association for Diabetes Education and Care (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: START-J; UMIN000004047 (Other: UMIN)
Record Dates: First submitted 2010-08-16; First posted 2010-08-17 (Estimated); Results first posted 2017-04-14 (Actual); Last update posted 2017-04-14 (Actual); Status verified 2017-03

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; Sitagliptin; Glimepiride; Elderly patients; Japanese
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; glimepiride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sitagliptin (Experimental)
  Interventions: Drug: Sitagliptin
- Glimepiride (Active Comparator)
  Interventions: Drug: Glimepiride

INTERVENTIONS:
Drug: Sitagliptin — Starting dose for sitagliptin is 50mg per day, can be increased up to 100mg (25-50mg; estimate glomerular filtration rate (eGFR) 30=< <50).
  Arms: Sitagliptin
Drug: Glimepiride — Starting dose for glimepiride is 0.5mg per day, can be increased up to 6.0mg
  Arms: Glimepiride

SUMMARY:
The purpose of this study is to compare the efficacy and the safety of sitagliptin and glimepiride in drug naïve elderly patients with Type 2 diabetes as evaluated by HbA1c change from baseline at 52 W as efficacy and incidence of hypoglycemia from randomization to 52 W as safety. The clinical hypotheses are non-inferiority of sitagliptin to glimepiride in efficacy as judged by HbA1c change from baseline at 52 W and superiority of sitagliptin to glimepiride in safety as judged by incidence of hypoglycemia in drug naïve elderly patients with T2DM. In addition, comparison of efficacy is extended to 104 W.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with type 2 diabetes who are oral hypoglycemic agent naive or, α-glucosidase inhibitor or biguanide monotherapy (to be washed out 4 weeks prior to randomization)
2. Signed informed consent obtained before any trial-related activities
3. Treatment with diet and exercise for 12 weeks and longer at screening
4. Age =>60 y.o.
5. Male and Female
6. HbA1c 6.9%=< <8.9%

Exclusion Criteria:

1. Active proliferative retinopathy or maculopathy requiring treatment
2. Liver dysfunction (>x2 of upper normal limit), moderate or severe renal dysfunction(serum Cr>1.5mg/dL in male, Cr>1.3mg/dL in female, eGFR<30), severe cardiac disease (NYHA III or IV), malignancy or uncontrolled hypertension (treated or untreated) as judged by the Investigator
3. Mental incapacity (including moderate or severe dementia) precluding adequate understanding and/or cooperation as judged by the Investigator
4. Recurrent hypoglycaemia or hypoglycaemic unawareness as judged by the investigator
5. Previous history of severe allergy to pharmaceutical products
6. Systemic glucocorticoids users or potential users
7. Suspected type 1 diabetes (including slowly progressive insulin dependent diabetes mellitus) or positive anti-glutamic acid decarboxylase antibody
8. Any condition that the investigator considers a potential obstacle to trial participation and/or data analysis

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2010-08; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yasuo Terauchi, M.D., Ph.D., Principal Investigator — Yokohama City University School of Medicine
Locations (1):
- Japan Association for Diabetes Education and Care, Chiyoda-Ku, Tokyo, Japan

REFERENCES:
- [Derived] Terauchi Y, Yamada Y, Ishida H, Ohsugi M, Kitaoka M, Satoh J, Yabe D, Shihara N, Seino Y. Efficacy and safety of sitagliptin as compared with glimepiride in Japanese patients with type 2 diabetes mellitus aged >/= 60 years (START-J trial). Diabetes Obes Metab. 2017 Aug;19(8):1188-1192. doi: 10.1111/dom.12933. Epub 2017 Apr 12. PMID 28294488
- See also: Related Info — https://www.nittokyo.or.jp/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sitagliptin | Glimepiride
Started | 153 | 152
Received Study Drug (Analysis set of evaluation for safety) | 148 | 143
Continued Treatment for 12 Weeks (Analysis set of evaluation for efficacy; Per Protocol Set) | 143 | 129
Completed 52-week Treatment | 119 | 111
Enrolled in Extension Study | 80 | 61
Completed (104-week extension study) | 76 | 60
Not Completed | 77 | 92
Not completed — Adverse Event | 8 | 6
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 14 | 7
Not completed — Physician Decision | 5 | 8
Not completed — Withdrawal by Subject | 6 | 11
Not completed — Nonparticipation in Extension Study | 39 | 50
Not completed — Did not receive study drug | 5 | 9

BASELINE CHARACTERISTICS:
Population: Analysis set of evaluation for efficacy ; Per Protocol Set
Groups:
- Sitagliptin: Starting dose for sitagliptin is 50mg per day, can be increased up to 100mg (25-50mg; eGFR 30=< <50).
- Total: Total of all reporting groups
Arm/Group | Sitagliptin | Glimepiride | Total
Number analyzed (Participants) | 143 | 129 | 272
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.2 (5.4) | 70.8 (5.5) | 70.5 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 50 | 119
  Male | 74 | 79 | 153
Region of Enrollment [Number; unit: participants]
  Japan | 143 | 129 | 272
HbA1c [Mean (Standard Deviation); unit: percent] | 7.48 (0.68) | 7.49 (0.67) | 7.48 (0.67)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 24.1 (3.3) | 24.2 (3.6) | 24.2 (3.4)
eGFR [Mean (Standard Deviation); unit: mL/min/1.73m^2] | 68.8 (17.1) | 67.9 (17.1) | 68.4 (17.1)
Body weight [Mean (Standard Deviation); unit: kg] | 60.9 (9.7) | 60.9 (9.7) | 60.9 (9.7)
HOMA-β [Mean (Standard Deviation); unit: percent] | 43.3 (33.7) | 38.5 (34.0) | 41.1 (33.9)
Insulin/Proinsulin Ratio [Mean (Standard Deviation); unit: ratio] | 0.217 (0.122) | 0.205 (0.129) | 0.211 (0.125)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c at 52 W
Time Frame: Baseline and 52 W
Population: Analysis set of evaluation for efficacy; Per Protocol Set.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent
Arm/Group | Sitagliptin | Glimepiride
Number analyzed (Participants) | 143 | 129
percent | -0.66 [-0.77 to -0.54] | -0.77 [-0.88 to -0.66]
Statistical Analysis 1: Comparison: Sitagliptin vs Glimepiride; Test type: Non-Inferiority or Equivalence — The pre-defined non-inferiority margin was 0.3%; p = 0.087, ANCOVA; LS mean difference = 0.11, 95% CI 2-sided [-0.02 to 0.24]

2. Primary Outcome: Number of Participants With Hypoglycaemia
Time Frame: From baseline to 52 W
Population: Analysis set of evaluation for safety.
Measure: Count of Participants; unit: Participants
Arm/Group | Sitagliptin | Glimepiride
Number analyzed (Participants) | 148 | 143
Participants | 7 | 23
Statistical Analysis 1: Comparison: Sitagliptin vs Glimepiride; Test type: Superiority or Other; p = 0.002, Fisher Exact

3. Secondary Outcome: The Number of Participants Achieving HbA1c < 6.9 %
Time Frame: 52 W
Population: Analysis set of evaluation for efficacy; Per Protocol Set Some participants were not completed to 52 W.
Measure: Count of Participants; unit: Participants
Arm/Group | Sitagliptin | Glimepiride
Number analyzed (Participants) | 134 | 128
Participants | 89 | 86
Statistical Analysis 1: Comparison: Sitagliptin vs Glimepiride; Test type: Superiority or Other; p = 1.0, Fisher Exact

4. Secondary Outcome: Change From Baseline in HOMA-β at 52 W
Description: β cell function is measured by the Homeostatic Model Assessment(HOMA-β). HOMA β = [20 x fasting insulin (μU/mL)] / [fasting plasma glucose (mmol/L) - 3.5]
Time Frame: Baseline and 52 W
Population: Analysis set of evaluation for efficacy; Per Protocol Set. Some participants had loss of the measurement.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Sitagliptin | Glimepiride
Number analyzed (Participants) | 122 | 119
percent | 10.2 (35.7) | 23.7 (56.1)
Statistical Analysis 1: Comparison: Sitagliptin vs Glimepiride; Test type: Superiority or Other; p = 0.030, ANCOVA

5. Secondary Outcome: Change From Baseline in Insulin/Proinsulin Ratio at 52 W
Time Frame: Baseline and 52 W
Population: Analysis set of evaluation for efficacy; Per Protocol Set. Some participants had loss of the measurement.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Sitagliptin | Glimepiride
Number analyzed (Participants) | 120 | 112
ratio | -0.049 (0.111) | -0.002 (0.095)
Statistical Analysis 1: Comparison: Sitagliptin vs Glimepiride; Test type: Superiority or Other; p < 0.001, ANCOVA

6. Secondary Outcome: Change From Baseline in Body Weight at 52 W
Time Frame: Baseline and 52 W
Population: Analysis set of evaluation for efficacy; Per Protocol Set. Some participants had loss of the measurement.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Sitagliptin | Glimepiride
Number analyzed (Participants) | 134 | 127
kg | -0.367 (2.441) | 0.309 (2.915)
Statistical Analysis 1: Comparison: Sitagliptin vs Glimepiride; Test type: Superiority or Other; p = 0.043, ANCOVA

ADVERSE EVENTS:
Arm/Group | Sitagliptin | Glimepiride
Serious Adverse Events (participants affected / at risk) | 13/148 | 3/143
Other Adverse Events (participants affected / at risk) | 33/148 | 31/143
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sitagliptin (N=148) | Glimepiride (N=143)
Pneumonia (Infections and infestations) | 1 | 0
Infectious enteritis (Infections and infestations) | 1 | 0
Acute myeloid leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hemorrhagic diathesis (Blood and lymphatic system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Hyphema (Eye disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Complete atrioventricular block (Cardiac disorders) | 0 | 1
Takotsubo cardiomyopathy (Cardiac disorders) | 1 | 0
Colon polyp (Gastrointestinal disorders) | 0 | 1
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Death (General disorders) | 0 | 1
Globe rupture (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sitagliptin (N=148) | Glimepiride (N=143)
Intestinal abscess (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 2 | 0
Cystitis (Infections and infestations) | 3 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 8 | 7
Pharyngitis (Infections and infestations) | 1 | 0
Helicobacter infection (Infections and infestations) | 0 | 1
Bile ｄuct ｃancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon ｃancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Polycythemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0
Mediastinal lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 2
Loss of appetite (Metabolism and nutrition disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Hypoesthesia (Nervous system disorders) | 0 | 2
Loss of consciousness (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 1 | 0
Allergic conjunctivitis (Eye disorders) | 0 | 1
Pterygium (Eye disorders) | 0 | 1
Retinal hemorrhages (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Heart failure (Cardiac disorders) | 0 | 1
Myocardial ischemia (Cardiac disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Erosive gastritis (Gastrointestinal disorders) | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Hemorrhoid (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Choledocholith (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Liver Cyst (Hepatobiliary disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Seborrheic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Hives (Skin and subcutaneous tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spondylosis deformans (Musculoskeletal and connective tissue disorders) | 1 | 0
Hygroma (Musculoskeletal and connective tissue disorders) | 0 | 1
Tenovaginitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Ureteral calculus (Renal and urinary disorders) | 0 | 1
Face edema (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 1
Fever (General disorders) | 0 | 1
Blood pressure increased (Investigations) | 0 | 1
Blood uric acid increased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
T-wave abnormality (Investigations) | 0 | 1
Injury (Injury, poisoning and procedural complications) | 2 | 0
Sprained ligament (Injury, poisoning and procedural complications) | 1 | 0
Wrist join fraction (Injury, poisoning and procedural complications) | 1 | 0
Ureteral stone removal (Surgical and medical procedures) | 0 | 1
Dental care (Surgical and medical procedures) | 1 | 0
Cataract operation (Surgical and medical procedures) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No